CLINICAL TRIAL: NCT01971008
Title: Abdominal Binders for the Treatment of Orthostatic Hypotension in Parkinson's Disease: an Investigator-initiated Randomized, Placebo-controlled, Cross-over Study
Brief Title: Abdominal Binder to Treat Orthostatic Hypotension (OH) in Parkinson's Disease (PD)
Acronym: ABOHP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Principal Investigator, Klaus Seppi, MD, Univ. Prof. Dr., Medical University Innsbruck
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: ABOHP
Record Dates: First submitted 2013-10-17; First posted 2013-10-28 (Estimated); Results first posted 2023-03-10 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2022-06

CONDITIONS: Parkinson's Disease; Neurogenic Orthostatic Hypotension in Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: N/A (the Intervention type in the present study was an elastic abdominal binder, which is a medical device)
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Elastic abdominal binder, then placebo binder (Experimental): Patients in this arm will be invited to wear an elastic abdominal binder ("Abdosyncro" Abdominalbandage, Syncro Med GmbH) for 2 hours on day 1 and a placebo binder ("Clima Care" Body warmer, Bort Medical) for 2 hours on day 3, after wash-out on day 2
  Interventions: Device: Elastic abdominal binder
- Placebo binder, then elastic abdominal binder (Experimental): Patients in this arm will be invited to wear a placebo binder ("Clima Care" Body warmer, Bort Medical) for 2 hours on day 1 and an elastic abdominal binder ("Abdosyncro" Abdominalbandage, Syncro Med GmbH) for 2 hours on day 3, after wash-out on day 2
  Interventions: Device: Placebo binder

INTERVENTIONS:
Device: Elastic abdominal binder
  Other Names: "Abdosyncro" Abdominalbandage, Syncro Med GmbH
  Arms: Elastic abdominal binder, then placebo binder
Device: Placebo binder
  Other Names: "Clima Care" Body warmer, Bort Medical
  Arms: Placebo binder, then elastic abdominal binder

SUMMARY:
The purpose of the present study is to determine whether the use of an abdominal binder is effective in the non-pharmacological management of orthostatic hypotension in patients suffering from Parkinson's disease

DETAILED DESCRIPTION:
In the present single blinded cross-over trial we investigated the effects of an elastic abdominal binder on blood pressure changes (systolic, diastolic and mean blood pressure) after 3 minutes of head-up tilt test in patients with Parkinson's disease and orthostatic hypotension.

Secondarily, we investigated the effects of an elastic abdominal binder on symptoms of orthostatic hypotension in daily living in a 4-weeks open-label follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic PD
* Hoehn & Yahr stadium < or = 4
* Age: 40-90
* Laboratory confirmed neurogenic orthostatic hypotension (NOH)
* Stable pharmacological therapy in the last 6 weeks
* Full legal competence

Exclusion Criteria:

* Other major neurologic or psychiatric diseases
* Untreated diabetes mellitus with clinical features of peripheral neuropathy
* Major cardiac diseases (ischemic, structural, arrhythmias)
* Evidence of varices (venous insufficiency stage > or = C2, "varicose veins")
* Known or suspected pregnancy
* Breast feeding

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-05; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Seppi, Univ. Prof. Dr., Principal Investigator — Department of Neurology - Medical University Innsbruck
Locations (1):
- Department of Neurology - Medical University Innsbruck, Innsbruck, Tyrol, Austria

REFERENCES:
- [Background] Seppi K, Weintraub D, Coelho M, Perez-Lloret S, Fox SH, Katzenschlager R, Hametner EM, Poewe W, Rascol O, Goetz CG, Sampaio C. The Movement Disorder Society Evidence-Based Medicine Review Update: Treatments for the non-motor symptoms of Parkinson's disease. Mov Disord. 2011 Oct;26 Suppl 3(0 3):S42-80. doi: 10.1002/mds.23884. PMID 22021174
- [Background] Ferreira JJ, Katzenschlager R, Bloem BR, Bonuccelli U, Burn D, Deuschl G, Dietrichs E, Fabbrini G, Friedman A, Kanovsky P, Kostic V, Nieuwboer A, Odin P, Poewe W, Rascol O, Sampaio C, Schupbach M, Tolosa E, Trenkwalder C, Schapira A, Berardelli A, Oertel WH. Summary of the recommendations of the EFNS/MDS-ES review on therapeutic management of Parkinson's disease. Eur J Neurol. 2013 Jan;20(1):5-15. doi: 10.1111/j.1468-1331.2012.03866.x. PMID 23279439
- [Background] Zesiewicz TA, Sullivan KL, Arnulf I, Chaudhuri KR, Morgan JC, Gronseth GS, Miyasaki J, Iverson DJ, Weiner WJ; Quality Standards Subcommittee of the American Academy of Neurology. Practice Parameter: treatment of nonmotor symptoms of Parkinson disease [RETIRED]: report of the Quality Standards Subcommittee of the American Academy of Neurology. Neurology. 2010 Mar 16;74(11):924-31. doi: 10.1212/WNL.0b013e3181d55f24. PMID 20231670
- See also: Coordination center for clinical studies of the Medical University Innsbruck — https://www.i-med.ac.at/kks/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 18 patients were screened for elegibility between May 2013 and January 2014 at the Department of Neurology of the Medical University of Innsbruck
Pre-assignment Details: 15 patients were randomized to receive either the abdominal binder or the Placebo binder first; 3 patients failed to meet all inclusion criteria.
Period: Overall Study
Arm/Group | Elastic Abdominal Binder, Then Placebo Binder | Placebo Binder, Then Elastic Abdominal Binder
Started | 6 | 9
Completed | 4 | 8
Not Completed | 2 | 1
Not completed — Protocol Violation | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Elastic Abdominal Binder, Then Placebo Binder | Placebo Binder, Then Elastic Abdominal Binder | Total
Number analyzed (Participants) | 6 | 9 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 4 | 8 | 12
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 69 [66 to 75] | 69 [66 to 75] | 69 [66 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 2 | 7 | 9
Region of Enrollment [Number; unit: participants]
  Austria | 12 | 12 | 12

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Blood Pressure (mmHg) After 3 Minutes of Passive Orthostatic Challenge From Baseline, When Wearing an Elastic Abdominal Binder vs a Placebo Binder for 2 Hours Each in People With Parkinson's Disease and Neurogenic Orthostatic Hypotension
Description: Using a single-blinded placebo-controlled cross-over design, 15 consecutive patients with PD and symptomatic OH were randomly assigned to first receive either an elastic abdominal binder (20±2mmHg pressure on the abdominal wall, Abdo-Syncro 3-stripes abdominal binder, Syncro Med GmbH) or a placebo binder (3±2mmHg pressure on the abdominal wall, Clima Care body warmer, Bort Medical GmbH) on two different days, separated by an interval of one day, to compare their efficacy on tilt-test examinations. On study day-1, all patients underwent a 1st baseline tilt-test examination. Afterwards they were asked to wear the assigned binder. Two hours later, the 1st study tilt-test was performed. The binder was subsequently taken off. Following interval on day-2, on study day-3 patients were crossed over to the other type of binder and underwent the same protocol as on day-1. Mean blood pressure was calculated as: (diastolic blood pressure +1/3(systolic blood pressure - diastolic blood pressure).
Time Frame: 3 days
Population: Fifteen patients were randomized. Three patients dropped-out during the cross-over phase (1 from the placebo-abdominal binder group and 2 from the abdominal binder-placebo group) and data from 12 patients were available for the primary outcome analysis.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Placebo Binder: Patients in this arm will be invited to wear a placebo binder ("Clima Care" Body warmer, Bort Medical) for 2 hours
  Placebo binder
- Elastic Abdominal Binder: Patients in this arm will be invited to wear an elastic abdominal binder ("Abdosyncro" Abdominalbandage, Syncro Med GmbH) for 2 hours
  Elastic abdominal binder
Arm/Group | Placebo Binder | Elastic Abdominal Binder
Number analyzed (Participants) | 12 | 12
mmHg | -2.3 (9.6) | 7.7 (6.6)

2. Secondary Outcome: Change in Systolic Blood Pressure (mmHg) After 3 Minutes of Passive Orthostatic Challenge From Baseline When Wearing an Elastic Abdominal Binder vs a Placebo Binder for 2 Hours Each in People With Parkinson's Disease and Neurogenic Orthostatic Hypotension
Description: Using a single-blinded placebo-controlled cross-over design, 15 consecutive patients with PD and symptomatic OH were randomly assigned to first receive either an elastic abdominal binder (20±2mmHg pressure on the abdominal wall, Abdo-Syncro 3-stripes abdominal binder, Syncro Med GmbH) or a placebo binder (3±2mmHg pressure on the abdominal wall, Clima Care body warmer, Bort Medical GmbH) on two different days, separated by an interval of one day, to compare their efficacy on tilt-test examinations. On study day-1, all patients underwent a 1st baseline tilt-test examination. Afterwards they were asked to wear the assigned binder. Two hours later, the 1st study tilt-test was performed. The binder was subsequently taken off. Following interval on day-2, on study day-3 patients were crossed over to the other type of binder and underwent the same protocol as on day-1.
Time Frame: 3 days
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo Binder | Elastic Abdominal Binder
Number analyzed (Participants) | 12 | 12
mmHg | -6.2 (14.7) | 9.3 (5.6)

3. Secondary Outcome: Change in Diastolic Blood Pressure (mmHg) After 3 Minutes of Passive Orthostatic Challenge From Baseline if Wearing an Elastic Abdominal Binder vs a Placebo Binder for 2 Hours Each in People With Parkinson's Disease and Neurogenic Orthostatic Hypotension
Description: as for outcome 2
Time Frame: 3 days
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Placebo Binder: Patients in this arm will be invited to wear a placebo binder ("Clima Care" Body warmer, Bort Medical) for 2 hours
- Elastic Abdominal Binder: Patients in this arm will be invited to wear an elastic abdominal binder ("Abdosyncro" Abdominalbandage, Syncro Med GmbH) for 2 hours
Arm/Group | Placebo Binder | Elastic Abdominal Binder
Number analyzed (Participants) | 12 | 12
mmHg | -0.3 (8.2) | 6.9 (8.2)

4. Secondary Outcome: Change in Mean Blood Pressure (mmHg) After 3 Minutes of Active Orthostatic Challenge From Baseline When Wearing an Elastic Abdominal Binder Versus a Placebo Binder for 2 Hours Each in People With Parkinson's Disease and Neurogenic Orthostatic Hypotension
Description: as for outcome 1
Time Frame: 3 days
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo Binder | Elastic Abdominal Binder
Number analyzed (Participants) | 10 | 10
mmHg | -6.4 (12.8) | 6.5 (7.9)

5. Secondary Outcome: Change in Supine Mean Blood Pressure (mmHg) if Wearing an Elastic Abdominal Binder vs a Placebo Binder for 2 Hours Each in People With Parkinson's Disease and Neurogenic Orthostatic Hypotension
Description: as for outcome 1
Time Frame: 3 days
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo Binder | Elastic Abdominal Binder
Number analyzed (Participants) | 12 | 12
mmHg | -2.2 (12.8) | 2.6 (13.7)

6. Secondary Outcome: Change in Orthostatic Hypotension Questionnaire Total Score After 4-weeks Open Label Trial With an Elastic Abdominal Binder With Respect to Baseline in People With Parkinson's Disease and Neurogenic Orthostatic Hypotension
Description: Upon completion of the single-blinded cross-over phase, patients were invited to wear the elastic abdominal binder on daily basis for 4 weeks. We evaluated the changes in the total score of the Orthostatic Hypotension Questionnaire (OHQ, which quantifies the impact of orthostatic symptoms in daily life) after these 4 weeks with respect to baseline. The OHQ is a 10-items scale. For each item the minimum score is 0 (no symptoms) and the max score is 10 (worst symptoms severity). The OHQ total score is calculated as follows: sum of the scores in each item/10 (total score range: 0-10). Higher values indicate worse outcomes.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: points (scale 0 to 10)
Groups:
- Open Label: All patients were invited to wear the elastic abdominal binder in a open label fashion
Arm/Group | Open Label
Number analyzed (Participants) | 12
points (scale 0 to 10) | -2.5 (1.5)

ADVERSE EVENTS:
Time Frame: 3 days (for the randomized, cross-over, single blinded phase) plus 4 weeks open label extension phase
Groups:
- Elastic Abdominal Binder: 3 days (cross-over phase) plus 4-weeks open-label extention phase
- Placebo Binder: 3 days (cross-over phase)
Arm/Group | Elastic Abdominal Binder | Placebo Binder
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/12
Other Adverse Events (participants affected / at risk) | 1/13 | 0/12
OTHER ADVERSE EVENTS (reported when occurring in more than 0.06% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Elastic Abdominal Binder (N=13) | Placebo Binder (N=12)
Gastro-esophageal reflux (Gastrointestinal disorders) | 1 (1) | NA — One patient reported exacerbation of gastroesophageal reflux during the 4-weeks open-label follow-up: this might have been related to regular use of the abdominal binder.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes